CLINICAL TRIAL: NCT06668844
Title: Endoscopic Direct "Draf IIa" (Carolyn's Window Approach) Versus Endoscopic Angled "Draf IIa"Approach in Chronic Rhinosinusitis With Frontal Sinus Affection ( A Comparative Study ).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hazem Gamal Noreldein, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Endoscopic direct Draf IIa
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Chronic Rhinosinusitis (CRS); Frontal Sinusitis; Draf I or IIa; Functional Endoscopic Sinus Surgery (FESS)
Keywords: Frontal sinusitis; Direct Draf; Endoscopic sinus surgery
MeSH Terms: conditions — Frontal Sinusitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First arm (Experimental): Endoscopic direct Draf IIa (Carolyn' window approach) frontal sinusotomy
  Interventions: Procedure: Endoscopic direct Draf IIa
- Second arm (Active Comparator): Endoscopic angled Draf IIa frontal sinuaotomy
  Interventions: Procedure: Endoscopic angled Draf IIa

INTERVENTIONS:
Procedure: Endoscopic direct Draf IIa — Endoscopic direct Draf IIa (Carolyn' window approach) frontal sinusotomy
  Arms: First arm
Procedure: Endoscopic angled Draf IIa — Group BFrontal sinusotomy using angled endoscopeand instruments
  Arms: Second arm

SUMMARY:
Patients with chronic rhinosinusitis with frontal sinus affection indicated for sinuscopy will be randomly categorized in 2 groups: group A will have endoscopic directDraf IIa frontal sinusotomy and group B will have endoscopic angled Draf IIa frontal sinusotomy, the two groups will be compared according to ostium patency and perioperative morbidity

DETAILED DESCRIPTION:
Frontal sinus surgery is a challenging component of endoscopic sinus surgery due to the intricacy and variability of frontal recess and sinus anatomy. Before the introduction of endoscopy in sinus surgery, complex cases of the frontal sinus were managed through the anterior wall using an osteoplastic flap approach. This technique was relatively successful in treating frontal sinus pathologies, but was invasive with adverse effects and failure in 6-25 percent of patients.

Different endoscopic techniques have been introduced for performing frontal sinusotomy. Draf categorized them into four techniques (Draf I, Draf IIa, Draf IIb, Draf III). Draf II procedures widen the frontal sinus outflow tract from the lamina papyracea laterally to the middle turbinate (Draf IIa) or the nasal septum medially (Draf IIb).

The thickness of the nasofrontal beak, and a limited anterior-posterior dimension of the frontal recess, make the Draf IIa frontal sinus surgery with angled endoscopy and instrumentation visually diffcult and requires skilled dexterity.

The direct access or Carolyn's window approach to the frontal recess replicates Draf's technique via the endoscopic approach. The approach utilizes only the 0° endoscope. In this approach, the entire frontal process of the maxilla, agger nasi and nasal process of the frontal bone, is removed with a high-speed drill.The goal of the approach is to visualize all walls of the frontal sinus via a ° endoscope. This postoperative view predicts better irrigation access and drainage of the frontal sinuses.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged 18 and above) with chronic rhino sinusitis affecting the frontal sinus with or without nasal polyps confirmed by nasal endoscopy and CT scan.
2. Unilateral or bilateral cases.
3. Denovo or recurrent cases.

Exclusion Criteria:

1. Individuals younger than 18 year-old.
2. Neoplasms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Assess endoscopic direct access Draf IIa (carolyn's window approach) in creating patent frontal sinusotomy. | 2 years
  Assess endoscopic direct access Draf IIa (carolyn's window approach) in creating patent frontal sinusotomy assessment will be done radiologically after 6 months : it will be considered patent if ostium more than 5mm

SECONDARY OUTCOMES:
Assess perioperative morbidity of endoscopic direct Draf IIa approach compared to endoscopic Draf IIa frontal sinusotomy with an angled endoscope and instrumentation | 2 years
  Assess perioperative morbidity of endoscopic direct Draf IIa approach compared to endoscopic Draf IIa frontal sinusotomy with an angled endoscope and instrumentation Defined as early (< 90 days) or late (> 90 days). Early morbidity: including
  1. bleeding (requiring intervention)
  2. pain (requiring additional analgesia)
  3. crusting (requiring additional post-op visit)
  4. adhesions (any)
  5. cerebrospinal fluid leak
  6. periorbital edema or hematoma
  7. inferior-based lateral wall mucosal flap necrosis. Late morbidity: including epiphora and smell reduction from baseline.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Barham HP, Hall CA, Hernandez SC, Zylicz HE, Stevenson MM, Zito BA, Harvey RJ. Impact of Draf III, Draf IIb, and Draf IIa frontal sinus surgery on nasal irrigation distribution. Int Forum Allergy Rhinol. 2020 Jan;10(1):49-52. doi: 10.1002/alr.22447. Epub 2019 Dec 11. PMID 31826329
- [Background] Spielman DB, Kim M, Overdevest J, Gudis DA. Zero-Degree Endoscopic Visualization of the Frontal Sinus Predicts Improved Topical Irrigation Delivery. Laryngoscope. 2021 Feb;131(2):250-254. doi: 10.1002/lary.28654. Epub 2020 Apr 11. PMID 32277702
- [Background] Seresirikachorn K, Sit A, Png LH, Kalish L, Campbell RG, Alvarado R, Harvey RJ. Carolyn's Window Approach to Unilateral Frontal Sinus Surgery. Laryngoscope. 2023 Oct;133(10):2496-2501. doi: 10.1002/lary.30569. Epub 2023 Jan 18. PMID 36651461
- [Background] Weber R, Draf W, Kratzsch B, Hosemann W, Schaefer SD. Modern concepts of frontal sinus surgery. Laryngoscope. 2001 Jan;111(1):137-46. doi: 10.1097/00005537-200101000-00024. PMID 11192882
- [Background] Hajbeygi M, Nadjafi A, Amali A, Saedi B, Sadrehosseini SM. Frontal Sinus Patency after Extended Frontal Sinusotomy Type III. Iran J Otorhinolaryngol. 2016 Sep;28(88):337-343. PMID 27738610
- [Background] Pagella F, Maiorano E, Turri-Zanoni M, Ferrari M, Carena P, Zoia C, Czaczkes C, Conti C, Schreiber A, Battaglia P, Emanuelli E, Pelucchi S, Bignami M, Nicolai P, Castelnuovo P. The role of the osteoplastic flap in the endoscopic era: a retrospective multicentre experience on revision surgery. Acta Otorhinolaryngol Ital. 2023 Apr;43(Suppl. 1):S34-S40. doi: 10.14639/0392-100X-suppl.1-43-2023-04. PMID 37698098
- [Background] Wormald PJ, Bassiouni A, Callejas CA, Kennedy DW, Citardi MJ, Smith TL, Orlandi RR, Kaschke O, Siow JK, Szczygielski K, Lund V, Fokkens W, Psaltis AJ. The International Classification of the radiological Complexity (ICC) of frontal recess and frontal sinus. Int Forum Allergy Rhinol. 2017 Apr;7(4):332-337. doi: 10.1002/alr.21893. Epub 2016 Dec 5. PMID 27918154